CLINICAL TRIAL: NCT00283673
Title: Impact of Aerobic Exercise Training on Age Related Changes in Insulin Sensitivity and Muscle Oxidative Capacity
Brief Title: Effect of Exercise Intervention on Various Physiologic Factors That Change With Increasing Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 350-95; R01AG009531 (NIH)
Record Dates: First submitted 2006-01-27; First posted 2006-01-30 (Estimated); Last update posted 2011-06-06 (Estimated); Status verified 2011-06

CONDITIONS: Aging
MeSH Terms: interventions — Exercise

INTERVENTIONS:
Behavioral: Exercise

SUMMARY:
This study randomized healthy sedentary people age 20-80 years to 16 weeks of supervised exercise versus no exercise. Several end points were evaluated after 16 weeks including insulin sensitivity and muscle physiology.

DETAILED DESCRIPTION:
Healthy subjects performing < 30 min exercise twice per week were studied prior to randomization and after of sixteen weeks exercise. They were randomized to sixteen weeks of supervised exercise performed on a stationary bike vs. placebo exercise (a series of flexibility exercises performed at home). Intensity, duration and frequency of exercise were gradually increased to four sessions per week lasting forty minutes each and achieving 80% target heart rate. Participants were weighed perioidically and counseled appropriately when weight changed by > 2 %. Insulin sensitivity and muscle mitochondrial protein synthesis were studied.

ELIGIBILITY:
Healthy subjects performing < 30 min exercise twice per week. Age 20-90 years. Willing to be randomized to exercise versus no exercise. Willing to be studied in General Clinical Research Center with studies including Muscle Biopsy.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102
Dates: Start 1995-09; Primary Completion 1998-01 (Actual); Study Completion 1998-01 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity

SECONDARY OUTCOMES:
Muscle Mitochondrial Protein Synthesis
mRNA of mitochondrial genes
mRNA of genes involved in mitochondrial biogenesis

CONTACTS AND LOCATIONS:
Overall Officials: K. Sreekumaran Nair, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Short KR, Vittone JL, Bigelow ML, Proctor DN, Rizza RA, Coenen-Schimke JM, Nair KS. Impact of aerobic exercise training on age-related changes in insulin sensitivity and muscle oxidative capacity. Diabetes. 2003 Aug;52(8):1888-96. doi: 10.2337/diabetes.52.8.1888. PMID 12882902